CLINICAL TRIAL: NCT02948790
Title: Auditory Nerve Monitoring Using Intra-cochlear Stimulation in Subjects With Acoustic Neuroma : Feasibility Study
Brief Title: Auditory Nerve Monitoring Using Intra-cochlear Stimulation in Subjects With Acoustic Neuroma
Acronym: NeuriStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PIC_05
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Hearing Loss, Cochlear; Neurinoma of the Acoustic Nerve
MeSH Terms: conditions — Hearing Loss, Sensorineural; Neuroma, Acoustic | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuristim (Experimental): Electrical stimulation with the Neuristim and auditory nerve electrical response measurements (wave V).
  Interventions: Device: Neuristim
- Digisonic SP EVO cochlear implant (Active Comparator): Electrical stimulation with the patient's cochlear implant and auditory nerve electrical response measurements (wave V).
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Neuristim — Stimulation at high, medium and low intensity on apical, medial and basal Neuristim electrode
  Arms: Neuristim
Device: Cochlear implant — Stimulation at high, medium and low intensity on apical, medial and basal Cochlear implant electrode
  Other Names: Digisonic SP EVO
  Arms: Digisonic SP EVO cochlear implant

SUMMARY:
The aim of this study is to assess the auditory nerve functionality with an intraoperative approach following a surgical removal of acoustic neuroma in patients with severe to profound sensorineural hearing disabilities.

DETAILED DESCRIPTION:
Whatever the acoustic neuroma treatments, the patient risks a hearing loss. The global strategy of hearing care aims to preserve the quality of life and patient hearing. For severe to profound hearing loss and anatomical auditory nerve preservation, the cochlear implant is put forward compared to the auditory brainstem implant. Indeed, cochlear implant provides better speech outcomes. If cochlear implantation is not possible or no benefit for the patient, the brainstem implant is the most widely used. The Neuristim device is used to investigate the auditory nerve integrity following neuroma surgery or on an affected auditory nerve. The Neuristim is an intra-cochlear stimulator used in an intraoperative way. The intra-cochlear electrodes provide an electrical stimulation to auditory nerve fibers, and auditory nerve response measurements to these electrical stimulation are recorded and evaluated to determine the auditory nerve functionality. The Neuristim is a device for helping surgeons to choose the most appropriate implantable solution. 2 groups of patients will be involved in this study:

* a group of 17 patients with an acoustic neuroma or a past neuroma surgically removed or acoustic neuroma not requiring a surgery and with severe to profound hearing loss candidate for a cochlear implant or a auditory brainstem depending on the auditory nerve functionality,
* a group of 17 patients with severe to profound hearing loss candidate for a cochlear implant.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Patient with an acoustic neuroma already surgically removed with associated hearing loss (experimental group),
* Patient with an acoustic neuroma programmed to be surgically removed and candidates for an implantable hearing rehabilitation solution (experimental group),
* Patient with an acoustic neuroma that not need to be removed and candidate for an implantable hearing rehabilitation solution (experimental group), or
* Typical patient candidate for a cochlear implant (control group)

Exclusion Criteria:

* Cochlea malformation, cochlea ossification
* Vulnerable subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Wave V latency | perioperatively

SECONDARY OUTCOMES:
Complications | perioperatively, 15 days postoperatively
Impedance measurement | perioperatively
ergonomics of the Neuristim | perioperatively
  satisfaction questionnaire
Speech audiometry | 3 months postoperatively
  in quiet and in noise
Pure tone audiometry | 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Vincent, MD, Principal Investigator — Hospital University Lille-Roger Salengro
Locations (4):
- France (4):
  - University Hospital Bordeaux - Pellegrin, Bordeaux
  - University Hospital Grenoble - A. Michallon, Grenoble
  - University Hospital Lyon - Edouard Herriot, Lyon
  - University Hospital Pitié Salpétrière, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: oticon medical website — http://www.oticonmedical.com